CLINICAL TRIAL: NCT06616948
Title: Examining the Reach, Effectiveness and Maintenance of Social Engagement on Exercise Outcomes: In-home Cycling for Individuals With Parkinson Disease
Brief Title: In-home Cycling for Individuals With PD: Effectiveness
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2018-0414: Effectiveness; A176000 (Other: UW Madison); EDUC\KINESIOLOGY\KINESIO (Other: UW Madison)
Record Dates: First submitted 2024-09-25; First posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Parkinson Disease
Keywords: social support; exercise
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Intervention Model Description: The proposed pilot study will utilize the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation and Maintenance) to focus on the reach and effectiveness of a 6-month triweekly in-home cycling program and then pilot a health coach model to promote maintenance for the subsequent 3-month period.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Social Cycling Group (Experimental): Exercise bike delivered to their home, custom fit to their needs and installed in a safe location, sessions will consist of up to 30 minutes of cycling while engaged in social interaction with a research staff member, thus providing a social/community aspect that would not otherwise be present.
  Interventions: Behavioral: Social Cycling Group
- Normal care control (No Intervention): Participants assigned to the normal care control will receive no intervention for the first 6-months then cross over to the cycling intervention.
- Biweekly health coach (Experimental): Following completion of the 6-month cycling intervention, participants will receive a call every 2-weeks to discuss ongoing maintenance efforts.
  Interventions: Behavioral: coaching calls
- No health coach (Active Comparator): Following the conclusion of the 6-month cycling session, participants will be contacted monthly to record falls. No discussion of ongoing exercise will occur
  Interventions: Behavioral: No coaching calls

INTERVENTIONS:
Behavioral: Social Cycling Group — engaged with a research staff member for 30 minutes of cycling
  Arms: Social Cycling Group
Behavioral: coaching calls — individuals will receive a phone call every 14 days to discuss ongoing exercise maintenance efforts.
  Arms: Biweekly health coach
Behavioral: No coaching calls — Following completion of the 6-month cycling sessions, no maintenance calls will be placed.
  Arms: No health coach

SUMMARY:
This study seeks to examine the reach and maintenance of an in-home cycling program for underserved individuals with Parkinson disease and to determine the effectiveness of a 6-month in-home, progressive, tele-exercise cycling program and 3-month health coach follow-up for those same participants.

DETAILED DESCRIPTION:
The benefits of exercise for individuals with Parkinson disease (PD) have been well documented; however, individuals with PD living in rural and underserved urban settings are largely unable or unwilling to participate in group exercise programs due in large part to their distance from such programs and financial considerations. Additionally, community based programs which provide social support and engagement have been shown to benefit elderly individuals as well as individuals with pathology, but are equally unattainable to this group. Taking the exercise to these individuals via telemedicine or tele-exercise may be an ideal means of delivering this type of intervention.

The long-term goal of this project is to improve outcomes for underserved populations of individuals with Parkinson disease (PD) by providing access to in-home physical activity via a telehealth approach. Approximately one million Americans currently live with a diagnosis of PD and it has been estimated that delaying the progression by 20% would result in a $75,891 savings per individual based on reduced health care costs, income maintenance, increased duration of life and improved quality of life. However, individuals with PD of lower socioeconomic status, people of color and rural dwelling seniors have been critically underserved by clinical and academic programming resulting in poorer health outcomes.

This study examines 1) the Reach, Effectiveness, Implementation and Maintenance and 2) the optimal delivery method for an in-home exercise intervention program for individuals with PD living in underserved communities. A managed and meaningful exercise intervention will be delivered that not only addresses the benefits of physical activity for individuals with PD, but also offers a social connection to research staff outside of the participant's typical caregiver(s).

SPECIFIC AIM 1: Examine the reach and maintenance of an in-home cycling program for underserved individuals with PD. Reach will be assessed by examining the demographic characteristics of the individuals enrolled and through the administration of a questionnaire on objective and subjective socioeconomic status to better understand their level of accessibility to services, perceived barriers and economic status. The investigators will also explore the implementation of a health coach to promote effective maintenance of the program after the 6-month intervention. Finally, two interviews will be conducted to better understand strengths and weakness of the program and to better address the needs of the participants in future studies.

* Hypothesis 1a: Demographic characteristics including race and socioeconomic status of the enrolled participants will not statistically differ from the characteristics of the state of WI.
* Hypothesis 1b: Feedback from participant interviews will inform future delivery of the in-home cycling program.

SPECIFIC AIM 2: Determine the effectiveness of a 6-month in-home, progressive, tele-exercise cycling program and 3-month health coach follow-up for underserved populations of individuals with PD.

* Hypothesis 2a: Participants will improve performance of activities of daily living from baseline to posttest. These effects will be maintained at 3-month follow-up.
* Hypothesis 2b: Participants will significantly improve measures of gait and balance performance and non- significantly improve fall rate from baseline to posttest. These effects will be maintained at 3-month follow-up in the group piloting implementation of a health coach, but not in solo follow-up group. Falls data will allow for effect size calculations for future applications.
* Hypothesis 2c: Activity level as measured by an activity monitor will increase from baseline to posttest. This effect will be maintained at 3-month follow-up in health coach group, but not in the solo group.

Study Design: 40 qualified individuals will be paired based on disease severity (score on subsection III of the UPDRS) and age and randomly assigned to either the cycling group or the normal care control group for 6 months. For those in the cycling group, participants will interact via Skype with study team members during all cycling sessions. This intervention will allow the individuals enrolled to participate in regular exercise and a community activity that promotes social support and engagement. The proposed pilot maintenance model for the 3-month period following the intervention will implement a health coach model with scheduled sessions every other week to discuss goals and motivation while decreasing the total contact time with the participant. Individuals in the normal care control group will crossover and complete the cycling intervention following the initial 6 months.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of idiopathic "definite PD" based upon established criteria
* vision at or corrected to 20/40 or better
* ability to independently ambulate for at least 10 minutes continuously
* no reported vestibular or neurological disease (stroke or muscle disease) beyond their diagnosed PD
* score of greater than or equal to 78 (no evidence of dementia) on the telephone adaptation of the modified mini-mental state exam
* English Speaking

Exclusion Criteria:

* contraindication for exercise
* history of muscular or orthopedic diagnosis
* inability to participate in the full duration of the study
* currently exercising for 20 or more minutes per week

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2025-07 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM) scores | baseline, post-test (~6-months), 3-month follow up (~9-months)
  The Canadian Occupational Performance Measure (COPM) will be administered to assess the participant's self-report of performance and satisfaction on a scale of 1 to 10 on self-selected occupational tasks. Performance and satisfaction scores range from 1 (lowest) to 10 (highest) for each identified item. The averages for each of the top three occupational tasks will be reported.

SECONDARY OUTCOMES:
Change in Pittsburgh Sleep Quality Index | baseline, post-test (~6-months), 3-month follow up (~9-months)
  The Pittsburgh Sleep Quality Index measures participant quality of sleep in each of 7 domains over the last month: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleep medication, and daytime dysfunction. The total possible range of scores is 0-21 with 0 indicating no difficulties and 21 indicating severe difficulties.
Change in Timed Up and Go Test | baseline, post-test (~6-months), 3-month follow up (~9-months)
  The Timed Up and Go Test measures the amount of time (in seconds) that it takes for the participant to stand, walk 3 meters away, and return to the seated position.
Change in Four Square Step Test | baseline, post-test (~6-months), 3-month follow up (~9-months)
  The Four Square Step Test measures the amount of time it takes to step forward, sideways, backward, sideways (and then in the reverse direction back to the start) through the quadrants of a square, stepping over canes that defines its boundaries.
Change in Fall Frequency | baseline, post-test (~6-months), 3-month follow up (~9-months)
  The Fall History Questionnaire is a 6-item survey that asks about Fall rate in the last 2 weeks, last month, last 6 months, the typical cause of a fall, and how the fear of falling may influence daily activities. The hypothesis is that Fall frequency will be improved in the socially engaged cycling group and not with those cycling alone.
Change in Standardized Gait Analysis: Gait Velocity | baseline, post-test (~6-months), 3-month follow up (~9-months)
  A portable electronic walkway, embedded with sensors, will be used to measure spatiotemporal variables including normalized gait velocity. Participants will begin at a starting point two meters from the mat, then walk toward and step onto the mat to continue walking until they achieve the stop line located two meters off of the opposite side of the mat. Data will be collected for forward preferred speed, backward preferred speed, forward fast, tandem and dual task gait. Each participant will complete five trials for each condition or a minimum of 40 steps
Change in Functional Gait Analysis: Gait Velocity | baseline, post-test (~6-months), 3-month follow up (~9-months)
  A portable electronic walkway, embedded with sensors, will be used to measure normalized gait velocity while participants complete a functional shopping task on the instrumented surface.
Change in mini-BESTest Score | baseline, post-test (~6-months), 3-month follow up (~9-months)
  The mini-BESTest will be used to assess balance. This 14-item, clinical battery is used to assess balance in four component areas (anticipatory transitions, postural response, sensory orientation and dynamic gait) and provides a single number summary of balance performance. Scores range from 0 to 28 with higher scores indicate higher function.
Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) | baseline, post-test (~6-months), 3-month follow up (~9-months)
  Movement Disorder Society Unified Parkinson Disease Rating Scale (MDS-UPDRS) assesses disease progress and clinical symptom presentation in four parts: I - Non-motor experience of daily living; II - Motor experience of daily living; III - Motor; and IV Motor complications. Scores range from 0 to 199, with 199 indicating most severe.

OTHER OUTCOMES:
Change in Free Locomotion Gait Analysis: Time | baseline, post-test (~6-months), 3-month follow up (~9-months)
  Participants will be asked to walk throughout the laboratory space and through nearby ground-floor hallways outside the laboratory, while wearing miniature wearable sensors to record their motion. Sensors record time, acceleration, angular velocity, magnetic field, air pressure (altitude), and optionally relative distance.
Change in Free Locomotion Gait Analysis: Acceleration | baseline, post-test (~6-months), 3-month follow up (~9-months)
  Participants will be asked to walk throughout the laboratory space and through nearby ground-floor hallways outside the laboratory, while wearing miniature wearable sensors to record their motion. Sensors record time, acceleration, angular velocity, magnetic field, air pressure (altitude), and optionally relative distance.
Change in Free Locomotion Gait Analysis: Angular Velocity | baseline, post-test (~6-months), 3-month follow up (~9-months)
  Participants will be asked to walk throughout the laboratory space and through nearby ground-floor hallways outside the laboratory, while wearing miniature wearable sensors to record their motion. Sensors record time, acceleration, angular velocity, magnetic field, air pressure (altitude), and optionally relative distance.
Change in Free Locomotion Gait Analysis: Relative Distance | baseline, post-test (~6-months), 3-month follow up (~9-months)
  Participants will be asked to walk throughout the laboratory space and through nearby ground-floor hallways outside the laboratory, while wearing miniature wearable sensors to record their motion. Sensors record time, acceleration, angular velocity, magnetic field, air pressure (altitude), and optionally relative distance.
Change in Activity Level Measured by Number of Steps Taken per day | baseline, post-test (~6-months), 3-month follow up (~9-months)
  The hypothesis is that activity level as measured by an activity monitor will increase from baseline to posttest. This effect will be maintained at 3-month follow-up in health coach group, but not in the solo group.

CONTACTS AND LOCATIONS:
Overall Officials: Kristen A Pickett, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes
Dr. Pickett will be responsible for deciding when/to whom to disseminate coded data, and will work with other researchers if necessary to confirm that they have proper IRB approval/etc., as necessary. Required UW-Madison IRB approval would be obtained prior to the release of any data.